CLINICAL TRIAL: NCT02608411
Title: TIvantinib as Maintenance Treatment in Extended Small-cell Lung Cancer (TIMES). Phase II Clinical Trial, Single Arm, Two Stage
Brief Title: TIvantinib as Maintenance Treatment in Extended Small-cell Lung Cancer (TIMES)
Acronym: TIMES
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety results (applied in METIV-HCC trial) have led early termination
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOV-SCLC-1-2014 TIMES; 2014-002497-37 (EudraCT Number)
Record Dates: First submitted 2015-11-10; First posted 2015-11-18 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma, Small Cell
MeSH Terms: conditions — Carcinoma, Small Cell | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ-197 (Experimental): ARQ-197 360 mg twice/day by mouth (PO), with meals, continuously as maintenance treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: ARQ197

INTERVENTIONS:
Drug: ARQ197
  Other Names: Tivantinib

SUMMARY:
This study aims to assess the role of MET inhibitors as maintenance treatment in adult patients with extensive stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed extensive-stage SCLC
* Disease control after the first line platinum/etoposide treatment
* ECOG performance status of 0 or 1
* Measurable disease according to RECIST Version 1.1 criteria
* Adequate bone marrow, liver, and renal function.
* Formalin Fixed Paraffin Embedded (FFPE) or frozen tumor tissue material must be available.
* Resolution of any toxic effects of prior therapy according to NCI CTCAE, v 4.0
* Full recovery from significant complications of the surgery
* If childbearing age, use of double-barrier contraceptive measures, oral or abstaining from sexual intercourse during the study and up to 90 days after the last dose of chemotherapy
* Negative pregnancy test within 72 hours prior to the initiation of study treatment, if of childbearing potential
* Signed informed consent prior to beginning protocol specific procedures
* Patients must be available for treatment and follow-up

Exclusion Criteria:

* Previous therapies with Tivantinib or other known c-MET inhibitor
* Radiotherapy for target lesions and major surgical procedure within 4 weeks, prior to the inclusion in the study
* Palliative radiotherapy within 2 weeks prior to the inclusion in the study
* History of malignancy in the past five years, excluding basal cell the cervix, prostate cancer with a value of prostate-specific antigen <0.2 ng / mL
* History of cardiac disease
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infections
* Pregnant or lactating women or childbearing/reproductive potential not using adequate contraception
* Need for breastfeeding during or within 12 weeks of completion of the study
* Gastrointestinal disorders that may interfere with the absorption of Tivantinib
* Inability or unwillingness to swallow the complete doses of Tivantinib
* Any known contraindication to treatment and other significant comorbid conditions which could jeopardize participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Approximately 48 months
  PFS will be assessed From the date of enrollment to the date of first documented disease progression or to the date of death from any cause or to the date of a new anti-cancer therapy, whichever occurs first. Patients without a PFS event at the time of analysis will be censored at the date of last assessment.

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 48 months
  The survival status will be assessed every 12 weeks (±14 days) until 48 months. Patients alive at the time of analysis will be censored at the date of last assessment.
Disease control rate (DCR) | Approximately 48 months
  The DCR will be defined as the percentage of patients with complete response (CR), partial response (PR) and stable disease (SD) at enrollment until the final visit
Occurrence of all grade toxicity events assessed by CTCAE v4.0 | Toxicity will be recorded during the treatment, until 30 days after the last dose of study medication, and graded according to the NCI- Common Terminology Criteria for Adverse Events (CTCAE) v.4.
  Toxicity will be analyzed in an "as treated" population, provided patients had received at least one dose of therapy.
Quality of Life | Approximately 48 months
  The instruments used for assessing the quality of life are the EORTC QLQ-C30 and QLQ-LC13 questionnaires. Quality of Life will be assessed from the date of enrollment until the end of treatment visit, that is anticipated after maximum 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Pasello, MD, Principal Investigator — Istituto Oncologico Veneto IRCCS
Locations (1):
- Istituto Oncologico Veneto, Padua, Italy